CLINICAL TRIAL: NCT06325605
Title: Medical Practitioner
Brief Title: Efficacy and Safety of Bifidobacterium Combined With High-frequency Transcranial Magnetic Stimulation in the Treatment of Adolescent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhen-Hong Hu (Other)
Responsible Party: Sponsor-Investigator, Zhen-Hong Hu, Associate chief physician, Tangshan Worker's Hospital
Organization: Tangshan Worker's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRYY-LL-KJ2022-064
Record Dates: First submitted 2024-03-04; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Adolescent Depression
MeSH Terms: interventions — Long-Term Synaptic Depression; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation group (Experimental): Patients in the observation group were treated with oral Bifidobacterium (0.07g/capsule, approval number: Guo Yao Zhun Zi S10950032, Shanghai Sine Pharmaceutical Co., Ltd.) 3 capsules, 3 times a day, for 8 consecutive weeks, and high-frequency rTMS. In the rTMS treatment, the transcranial magnetic stimulation device with an "8"-shaped coil with a diameter of 70mm was placed on the dorsolateral area of the left prefrontal lobe of the patient. The motor threshold was set to 90%. A 10-Hz pulse sequence was applied for 4 secs followed by a 20 secs interval. 10 pulses per train were used, and the total stimulation time was 30mins per day, 4 times a week, for 8 consecutive weeks.
  Interventions: Drug: Bifidobacterium; Device: High-frequency rTMS
- Control group (Active Comparator): Patients in the control group were treated with oral escitalopram oxalate (manufacturer: Sichuan Kelun Pharmaceutical Co., Ltd.; approval No.: Guo Yao Zhun Zi H20080788). The initial dose was 5mg/d, for 7 consecutive days. The dose was increased to 10 mg/d according to the tolerance of the patients for another 7 consecutive days, and then to 20 mg/d according to the patient's condition and tolerance for 8 weeks.
  Interventions: Drug: Escitalopram Oxalate

INTERVENTIONS:
Drug: Bifidobacterium — 3 capsules, 3 times a day, for 8 consecutive weeks
  Other Names: 0.07g/capsule, approval number: Guo Yao Zhun Zi S10950032, Shanghai Sine Pharmaceutical Co., Ltd.
  Arms: Observation group
Device: High-frequency rTMS — In the rTMS treatment, the transcranial magnetic stimulation device with an "8"-shaped coil with a diameter of 70mm was placed on the dorsolateral area of the left prefrontal lobe of the patient. The motor threshold was set to 90%. A 10-Hz pulse sequence was applied for 4 secs followed by a 20 secs interval. 10 pulses per train were used, and the total stimulation time was 30mins per day, 4 times a week, for 8 consecutive weeks.
  Arms: Observation group
Drug: Escitalopram Oxalate — Oral escitalopram oxalate. The initial dose was 5mg/d, for 7 consecutive days. The dose was increased to 10 mg/d according to the tolerance of the patients for another 7 consecutive days, and then to 20 mg/d according to the patient's condition and tolerance for 8 weeks
  Other Names: manufacturer: Sichuan Kelun Pharmaceutical Co., Ltd.; approval No.: Guo Yao Zhun Zi H20080788
  Arms: Control group

SUMMARY:
A total of 100 patients with adolescent depression who were admitted to our hospital between March 2022 and October 2022 were selected. On the basis of double blinding, these patients were randomly divided into the observation group(n=50) and the control group(n=50) using a random number table. 5S management method was used in the whole process of treatment to improve the hospital environment, increase the work efficiency and reduce the occurrence of cross infection through the effective implementation of the five steps of sort(Seiri), set in order(Seiton), shine (Seiso), standardize(Seiketsu) and sustain(Shitsuke).

ELIGIBILITY:
Inclusion Criteria:

* aged 13-18 years old;
* met the diagnostic criteria for depression in the International Classification of Disease-10 (ICD-10);
* with a total score of the Hamilton Rating Scale for Depression (HAMD-24) ≥20 in the initial assessment;
* who were right-handed

Exclusion Criteria:

* with a definite diagnosis of other mental disorders in the past;
* with a past or current history of manic episodes;
* with a past or current history of severe physical diseases;
* who used antidepressants, mood stabilizers, steroids, anti-inflammatory drugs, antibiotics, and immunomodulators in the past 1 month;
* who used lactic acid bacteria products for ≥7 days in the past 1 month;
* with a history of alcohol or psychoactive substance abuse within the last 3 months;
* with contraindications for rTMS, including but not limited to intracranial metal foreign bodies, cardiac pacemakers, and ear hearing aids;
* complicated with organic brain diseases, epileptic diseases, and severe physical diseases

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
HAMD-24 scores | 4 times a week, for 8 consecutive weeks
  Final scores were interpreted as no depression (<20), mild or moderate depression (≥20), and severe depression (≥35)
TNF-α | 7 consecutive days
  About 5ml of fasting venous blood was collected in the morning, centrifuged at 3000rpm for 10mins, and the upper serum was collected. The levels of serum tumor necrosis factor-α(TNF-α), interleukin-1β(IL-1β), IL-6, dopamine(DA), 5-hydroxytryptamine(5-HT) and cortisol(COR) were measured by ELISA using an automatic biochemical analyzer(Dxc800, Beckman, USA). The relative expression levels of serum miR-16 and miR-195 were determined by PCR. All measurements were strictly conducted by laboratory specialists following the instructions of the instruments and kits.
IL-1β | 7 consecutive days
  About 5ml of fasting venous blood was collected in the morning, centrifuged at 3000rpm for 10mins, and the upper serum was collected. The levels of serum tumor necrosis factor-α(TNF-α), interleukin-1β(IL-1β), IL-6, dopamine(DA), 5-hydroxytryptamine(5-HT) and cortisol(COR) were measured by ELISA using an automatic biochemical analyzer(Dxc800, Beckman, USA). The relative expression levels of serum miR-16 and miR-195 were determined by PCR. All measurements were strictly conducted by laboratory specialists following the instructions of the instruments and kits.
IL-6 | 7 consecutive days
  About 5ml of fasting venous blood was collected in the morning, centrifuged at 3000rpm for 10mins, and the upper serum was collected. The levels of serum tumor necrosis factor-α(TNF-α), interleukin-1β(IL-1β), IL-6, dopamine(DA), 5-hydroxytryptamine(5-HT) and cortisol(COR) were measured by ELISA using an automatic biochemical analyzer(Dxc800, Beckman, USA). The relative expression levels of serum miR-16 and miR-195 were determined by PCR. All measurements were strictly conducted by laboratory specialists following the instructions of the instruments and kits.
DA | 7 consecutive days
  About 5ml of fasting venous blood was collected in the morning, centrifuged at 3000rpm for 10mins, and the upper serum was collected. The levels of serum tumor necrosis factor-α(TNF-α), interleukin-1β(IL-1β), IL-6, dopamine(DA), 5-hydroxytryptamine(5-HT) and cortisol(COR) were measured by ELISA using an automatic biochemical analyzer(Dxc800, Beckman, USA). The relative expression levels of serum miR-16 and miR-195 were determined by PCR. All measurements were strictly conducted by laboratory specialists following the instructions of the instruments and kits.
5-HT | 7 consecutive days
  About 5ml of fasting venous blood was collected in the morning, centrifuged at 3000rpm for 10mins, and the upper serum was collected. The levels of serum tumor necrosis factor-α(TNF-α), interleukin-1β(IL-1β), IL-6, dopamine(DA), 5-hydroxytryptamine(5-HT) and cortisol(COR) were measured by ELISA using an automatic biochemical analyzer(Dxc800, Beckman, USA). The relative expression levels of serum miR-16 and miR-195 were determined by PCR. All measurements were strictly conducted by laboratory specialists following the instructions of the instruments and kits.
COR | 7 consecutive days
  About 5ml of fasting venous blood was collected in the morning, centrifuged at 3000rpm for 10mins, and the upper serum was collected. The levels of serum tumor necrosis factor-α(TNF-α), interleukin-1β(IL-1β), IL-6, dopamine(DA), 5-hydroxytryptamine(5-HT) and cortisol(COR) were measured by ELISA using an automatic biochemical analyzer(Dxc800, Beckman, USA). The relative expression levels of serum miR-16 and miR-195 were determined by PCR. All measurements were strictly conducted by laboratory specialists following the instructions of the instruments and kits.
Serum miR-16 | 7 consecutive days
  About 5ml of fasting venous blood was collected in the morning, centrifuged at 3000rpm for 10mins, and the upper serum was collected. The levels of serum tumor necrosis factor-α(TNF-α), interleukin-1β(IL-1β), IL-6, dopamine(DA), 5-hydroxytryptamine(5-HT) and cortisol(COR) were measured by ELISA using an automatic biochemical analyzer(Dxc800, Beckman, USA). The relative expression levels of serum miR-16 and miR-195 were determined by PCR. All measurements were strictly conducted by laboratory specialists following the instructions of the instruments and kits.
Serum miR-195 | 7 consecutive days
  About 5ml of fasting venous blood was collected in the morning, centrifuged at 3000rpm for 10mins, and the upper serum was collected. The levels of serum tumor necrosis factor-α(TNF-α), interleukin-1β(IL-1β), IL-6, dopamine(DA), 5-hydroxytryptamine(5-HT) and cortisol(COR) were measured by ELISA using an automatic biochemical analyzer(Dxc800, Beckman, USA). The relative expression levels of serum miR-16 and miR-195 were determined by PCR. All measurements were strictly conducted by laboratory specialists following the instructions of the instruments and kits.

CONTACTS AND LOCATIONS:
Locations (1):
- Tangshan Workers' Hospital, Tangshan, Hebei, China